CLINICAL TRIAL: NCT01081639
Title: Phase III Study on the Convenience, Safety and Efficacy of Follitropin Alfa Liquid Formulation Applied by a Pen Versus Follitropin Beta Liquid Formulation Applied by Pen
Brief Title: To Evaluate the Convenience, Safety and Efficacy of Follitropin Alfa Liquid Pen Compared With Follitropin Beta Liquid Pen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono GmbH, Germany (Industry)
Responsible Party: PD Dr. habil. Christoph Keck, Universitätsfrauenklinik, Hugstetter Straße 55, 79106 Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP 24554
Record Dates: First submitted 2010-02-22; First posted 2010-03-05 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2010-11

CONDITIONS: Infertility; Ovulation Induction
Keywords: Follitropin alfa; Follitropin beta; Fertilization, in vitro; Intracytoplasmic sperm injection; Assisted reproductive techniques; Polycystic ovary syndrome
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — follitropin alfa; follitropin beta

ARMS (2):
- Gonal-f (Experimental)
  Interventions: Drug: Follitropin alfa liquid formulation
- Puregon (Active Comparator)
  Interventions: Drug: Follitropin beta liquid formulation

INTERVENTIONS:
Drug: Follitropin alfa liquid formulation — Follitropin alfa (Gonal-f) liquid pen (300, 450 and 900 IU) was applied by subcutaneous (sc) administration. Regimen of recombinant FSH-stimulation followed the standard protocol of the IVF-center
  Other Names: Gonal-f
  Arms: Gonal-f
Drug: Follitropin beta liquid formulation — Follitropin beta (Puregon) liquid cartridge (300 and 600 IU) used with the Pen was applied by sc administration. Regimen of recombinant FSH-stimulation followed the standard protocol of the IVF-center
  Other Names: Puregon
  Arms: Puregon

SUMMARY:
This was a prospective, randomised, open comparative monocentric phase IIIb study to evaluate the convenience, safety and efficacy of follitropin alfa (Gonal-f) liquid pen compared with follitropin beta (Puregon) liquid pen.

DETAILED DESCRIPTION:
Treatment of subfertility and infertility by assisted reproduction technologies (ART) such as in-vitro fertilisation (IVF) and embryo transfer (ET) requires multiple follicular development to increase the number of female gametes, and the chances of a successful treatment outcome. Ovarian stimulation in IVF/intracytoplasmic sperm injection (ICSI) currently includes suppression of endogenous luteinizing hormone (LH) secretion by administration of a gonadotrophin releasing hormone (GnRH) agonist, followed by stimulation of multiple follicular development by exogenous FSH administration. When adequate follicular development is achieved, a single dose of u-hCG (urinary-hCG) is administered to mimic the endogenous LH surge and induce final oocyte maturation. Recombinant-human FSH (r-hFSH) has been shown to be superior to u-hFSH in terms of requiring fewer ampules and more efficacious in terms of number of oocytes recovered and in terms of pregnancy rates.

Recently, a new formulation of follitropin alfa has been developed due to a general trend in the field of therapeutic recombinant proteins to move from presentations based on biological activity to presentations based on physico-chemical characteristics. Until now follitropin alfa has been produced as a powder for injection (either as monodose or multidose preparations) in glass ampoules or in glass vials and administered using plastic or glass syringe. Serono developed a multidose solution for injection in a prefilled disposable injection pen. This study involved comparing the administration of follitropin alfa liquid formulation applied by pen with that of follitropin beta liquid formulation also applied by pen.

OBJECTIVES The objectives of this study were to evaluate the convenience, safety and efficacy of Follitropin alfa (Gonal-f) liquid pen compared with Follitropin beta (Puregon) liquid pen.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal woman, between her 18th and 39th birthday, receiving recombinant FSH as stimulation for IVF and/or ICSI
* Subjects who were able to communicate well with the investigator and to comply with the requirements of the entire study
* Subjects who had given written informed consent, prior to treatment, with the understanding that consent may be withdrawn by the subject at any time without prejudice

Exclusion Criteria:

* Subjects who had known allergic reaction against one of the ingredients
* Subjects with enlarged ovaries or cysts unrelated to polycystic ovaries (PCO)
* Subjects with gynaecological bleeding of unknown origin
* Subjects who had ovarian, uterine, or mammary cancer
* Subjects with tumors of the hypothalamus or the pituitary gland

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2003-11; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Convenience and Safety | 1 year
  Convenience parameters included nurse/subjects preference; time to train subject; operative tolerance and wastage of product which were assessed during the post-treatment period.
  Safety parameters included local reactions (pain, bruising, redness, itching, swelling)and adverse drug events which were assessed during the pre-treatment, treatment and post-treatment period.

SECONDARY OUTCOMES:
Efficacy | 1 year
  Collection of routine data from the RecDate registry such as: stimulation duration; FSH starting dose; FSH dosage on last treatment day; total amount of gonadotrophin needed; number of follicles on the day of the last ultra-scan; number of oocytes retrieved; number of fertilized oocytes; number of embryos transferred; wastage of product; number of cartridges of Gonal-f (300 IU, 450 IU, and 900 IU) and Puregon (300 IU and 600 IU) opened; clinical pregnancy by Ultra-scan (if already available at time point of final report writing).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Keck, PD, Dr. med., Principal Investigator — Universitätsfrauenklinik Freiburg

REFERENCES:
- [Result] Porter R, Kissel C, Saunders H, Keck C. Patient and nurse evaluation of recombinant human follicle-stimulating hormone administration methods: comparison of two follitropin injection pens. Curr Med Res Opin. 2008 Mar;24(3):727-35. doi: 10.1185/030079908X273291. Epub 2008 Jan 28. PMID 18230195